CLINICAL TRIAL: NCT06556524
Title: The Effect of Simulation Practice With a Live Subject on the Anxiety Level and Perceived Competence Level of Paramedic Candidates in Approaching a Trauma Patient
Brief Title: The Effect of Live Subject on the Anxiety Level and Perceived Competence Level
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sariye Bilge DOGAN, Lecturer, Gazi University
Other Study IDs: E-77082166-604.01.02-300721
Record Dates: First submitted 2024-08-06; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Anxiety Level
Keywords: Simulation; Paramedic; Anxiety; Competence
MeSH Terms: conditions — Anxiety Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- twenty four Group: vocational school students
  Interventions: Behavioral: observation

INTERVENTIONS:
Behavioral: observation — Behavioral observation and trauma measurement in live mannequin application

SUMMARY:
This study was carried out to examine the effect of training on the proficiency and anxiety levels of Paramedic students in a realistic, simulated environment of the pre-hospital scene. A total of 72 second-year students in the Paramedic program participated in this study with an interventional approach. The data collection form used in the study consisted of sociodemographic characteristics, a self-efficacy form for approaching trauma patients, and the worry and anxiety scale. Within the framework of the research, a competition named "trauma rally" was organized for university Paramedic students, which consisted of the pre-hospital approach of injured live subjects. Through face-to-face interviews, the data collection form was filled out with the participants before, immediately after and one month after the competition.

DETAILED DESCRIPTION:
Teaching-learning strategies are methods to make it easier for the student to achieve professional goals in personal development. In the context of the academic education of healthcare professionals, ethical issues, patient safety, technological developments, health science, complexity of care measurements and current business world necessities should be taken into account by considering these strategies. In this context, simulation-based learning is one of the most effective and interesting teaching strategies and has been shown to reduce gaps between education and practice and adapt nursing students to clinical environments. Simulation is a set of structured activities that represent actual or potential situations in training and practice. These activities allow participants to develop or increase their knowledge, skills and attitudes, or to analyze and respond to realistic situations in a simulated environment. Simulations are especially important in clinical environments because they imitate various aspects of the real world and provide safe learning environments where students can practice until they reach skill competence through self-correction. As a matter of fact, the European heart association (ERC) points out that simulation programs increase the quality of trauma and advanced life support training and increase resuscitation rates after cardiac arrest. High fidelity simulation-based training can be an important component in preparing students for a successful transition into clinical practice. Additionally, it contributes to student satisfaction, confidence, competence and reduced anxiety levels. For these reasons, simulated experiences may be an option to complement traditional healthcare professional education methods.

ELIGIBILITY:
Inclusion Criteria:

* volunteering

Exclusion Criteria:

* non volunteering

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: vocational school student
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
anxiety level and trauma cases | fifteen days
  As a result, it was determined that simulation training with a live subject did not change the anxiety level of paramedic candidates, but increased their self-efficacy against trauma cases, and that there was a negative relationship between anxiety scores and self-efficacy scores. Considering that interventions on patients and injured people in the pre-hospital scene are critical, it is recommended that simulation methods be combined with traditional methods in paramedic training.

CONTACTS AND LOCATIONS:
Overall Officials: Sariye Bilge Doğan, M.Sc, Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee BO, Liang HF, Chu TP, Hung CC. Effects of simulation-based learning on nursing student competences and clinical performance. Nurse Educ Pract. 2019 Nov;41:102646. doi: 10.1016/j.nepr.2019.102646. Epub 2019 Oct 23. PMID 31698255